CLINICAL TRIAL: NCT00616278
Title: National Cooperative Growth Study of Nutropin AQ, Nutropin, Protropin, and Nutropin Depot in Children With Growth Failure Due to Chronic Renal Insufficiency (CRI) or End-Stage Renal Disease (ESRD)
Brief Title: National Cooperative Growth Study in CKD
Acronym: NCGS
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200412150
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Failure AND; Chronic Renal Insufficiency OR; End Stage Renal Disease
MeSH Terms: conditions — Dwarfism, Pituitary; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn whether growth hormone being administered to children with Chronic Kidney Disease is effective and if it has any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient of the UC Davis Medical Center pediatric clinic with Chronic Kidney Disease

Exclusion Criteria:

* Greater than 18 years old
* Not a patient at the UC Davis Medical Center pediatric clinic

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures of the NCGS are ongoing safety and efficacy of Genentech GH preparations in pediatric growth disorders for which GH is initiated. | per the study, the pt will be on GH treatement until the physician instructs them to stop

CONTACTS AND LOCATIONS:
Overall Officials: Lavjay Butani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States